CLINICAL TRIAL: NCT01368484
Title: Effect of Dietary DHA Supplementation on Sperm Quality.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Valenciano de Infertilidad, IVI VALENCIA (Other)
Collaborators: University of Barcelona (Other)
Responsible Party: Juan Carlos Martínez Soto., Instituto Valenciano de infertilidad, Murcia, Spain.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IVI MUR 005-2009
Record Dates: First submitted 2011-06-07; First posted 2011-06-08 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2011-06

CONDITIONS: SPERM
MeSH Terms: interventions — Sunflower Oil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sunflower oil (Placebo Comparator)
  Interventions: Dietary Supplement: Sunflower oil
- Docosahexanoic acid (Experimental)
  Interventions: Dietary Supplement: Docosahexanoic acid

INTERVENTIONS:
Dietary Supplement: Sunflower oil — 1500 mg sunflower/day for 10 weeks
  Arms: Sunflower oil
Dietary Supplement: Docosahexanoic acid — 1500mg/day for 10 weeks
  Arms: Docosahexanoic acid

SUMMARY:
The aim of this study is evaluated the effect of dietetic supplementation with DHA on human sperm quality, antioxidant capacity and sperm DNA damage.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of male factor.

Exclusion Criteria:

* Metabolic and genetic diseases.
* Oncological patients.
* Patients with anticoagulants treatment.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2009-12; Primary Completion 2010-12 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
sperm concentration | 5 weeks
  million of spermatozoa per milimitre
Sperm motility | 5 weeks
  Percentage of motile sperm.
Sperm morphology | 5 weeks
  Percentage of sperm with normal morphology
Total capacity antioxidant | 5 weeks
  Total antioxidant capacity (TAC)is a colorimetric assay that measure the combined antioxidant activities of all its non enzymatic constituents in seminal plasma.
Sperm DNA damage. | 5 weeks
  DNA fragmentation analysis was evaluated by TUNEL test and measured by flow cytometry
Fatty acids measure. | 5 weeks
  Fatty acid analysis in seminal plasma and spermatozoa were evaluated by gas chromatography.The percentage of each fatty acid class was expressed as percentage of total fatty acids.

SECONDARY OUTCOMES:
Sperm in ejaculate | 5 weeks
  Million of spermatozoa in eyaculate.
Volume of ejaculate. | 5 weeks
  Eyaculated milliliters.
Sperm viability | 5 weeks
  Porcentage of sperm whitout membrane damage

CONTACTS AND LOCATIONS:
Overall Officials: Martinez Soto, Juan Carlos, Principal Investigator — IVI Murcia; Landeras Gutierrez, Jose, Study Director — IVI Murcia; Nicolas Arnau, Maria, Study Chair — IVI Murcia; Fernandez Olmedilla, Laura, Study Chair — IVI Murcia; Albero Pilar, Study Chair — IVI Murcia; Domingo JC, Study Chair — University of Barcelona
Locations (1):
- Instituto Valenciano de infertilidad, Murcia, Murcia, Spain